CLINICAL TRIAL: NCT02167919
Title: Efficacy of Prostatic Artery Embolization (PAE) in Patients With Severe Benign Prostatic Hyperplasia (BPH) As an Alternative to Open Prostatectomy
Brief Title: Efficacy of Prostatic Artery Embolization (PAE) in Patients With Severe Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 13-3445
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Prostate; Men; Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia; Multiple Endocrine Neoplasia Type 1; Hyperplasia | interventions — Microspheres

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prostatic artery embolization (Experimental): Microspheres measuring 100-300 microns will be injected under fluoroscopic guidance into the left and right prostatic arteries for embolization.
  Interventions: Device: Microspheres

INTERVENTIONS:
Device: Microspheres — Prostatic artery embolization (PAE) is a new procedure that decreases the size of the prostate by blocking its arterial blood flow. Through a tiny puncture in the upper thigh or forearm a catheter is directed to the prostatic artery using fluoroscopic guidance. Once in place, sub-millimeter particles are injected that obstruct the prostatic arteries resulting in gland ischemia, and ultimately, reduction in size. The technique has only been recently developed in Portugal and Brazil and has similarities to Uterine Artery Embolization used to treat uterine fibroids.

SUMMARY:
Purpose: To evaluate the efficacy of prostatic artery embolization (PAE) in patients with benign prostatic hyperplasia (BPH) and refractory lower urinary tract symptoms (LUTS) in decreasing the volume of the prostate gland.

Participants: Study participants will be recruited from UNC Urology clinics as well as referring providers. We will include 15 men who are experiencing LUTS not controlled by medication with estimated prostate gland weight between 80 and 150 grams.

Procedures (methods): Enrolled patients will undergo the standard work-up for a surgical prostate procedure. In addition, the patient's arteries will be evaluated with a pelvic CT angiogram. Then, patients will undergo prostatic artery embolization. Follow up visits will be scheduled at 1, 3, 6, and 12 months after the procedure.

At the end of the follow-up period, if reduction in prostate gland size has made the patient eligible for transurethral therapy, they may proceed to such procedure or elect to undergo no further surgical procedure, depending on residual symptoms. Similarly, if insufficient gland size reduction has occurred, the patient may elect to pursue OP or no further procedure if they are no longer bothered by LUTS.

DETAILED DESCRIPTION:
This will be an open label pilot study with a small population undergoing an intervention to determine safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age > 40
* Prostate gland measures between 80 and 150 grams
* Have previously taken BPH medication for 6 months without desired improvement of LUTS or has started medication and stopped due to unwanted side effects
* Moderate to severe LUTS as defined by IPSS score >18
* Peak urine flow rate (Qmax) <12 ml/sec
* Capable of giving informed consent
* Life expectancy greater than 1 year

Exclusion Criteria:

* Severe cardiac or pulmonary disease
* Uncontrolled diabetes mellitus
* Immunosuppression
* Neurogenic bladder and/or sphincter abnormalities secondary to Parkinson's disease, multiple sclerosis, cerebral vascular accident, diabetes, etc.
* Acute urinary retention
* Glomerular filtration rate less than 45 as approximated using using serum creatinine levels.
* Confirmed or suspected bladder cancer
* Recent (within 3 months) cystolithiasis or gross hematuria
* Urethral strictures, bladder neck contracture, or other potentially confounding bladder pathology
* Active urinary tract infection
* Previous rectal surgery or history of rectal disease if PAE, anoscopy or transrectal ultrasound are thought to potentially cause injury to the rectum due to the previous surgery or disease
* Previous pelvic radiation or radical pelvic surgery
* Confirmed or suspected malignancy of the prostate based on DRE, TRUS or PSA. (> 10 ng/ml or > 2.5 ng/ml and < 10 ng/ml with free PSA < 25% of total PSA without a negative biopsy)
* Uncorrectable coagulopathy including INR > 2.5 or platelets < 30,000

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Prostate size (grams) | 1 year
  Reduction in size of the prostate to less than 80 grams
Lower urinary symptoms (Arbitrary units) | 1 year
  Improvement of LUTS as defined by IPSS score <18.

SECONDARY OUTCOMES:
Procedure completion without complication (percentage) | 1 year
  Completion of PAE without major complication
Sexual Function (Arbitrary units) | 1 year
  Stability or improvement of sexual function as determined by an unchanged or improved score on the International Index of Erectile Function (IIEF) questionnaire
Quality of Life (Arbitrary units) | 1 year
  Improvement of quality of life as determined by an improved score on Quality of Life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ari Isaacson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No